CLINICAL TRIAL: NCT06642142
Title: Evaluation of the Onset and the Extent of Sensory Block After Thoracic ESP Block in Breast Surgery - a Prospective Observational Study
Brief Title: Onset of Sensory Block After Thoracic ESP Block
Status: Recruiting | Type: Observational
Sponsor: Ospedale Santa Maria Goretti (Other)
Responsible Party: Principal Investigator, Irene Lupelli, Doctor, Ospedale Santa Maria Goretti
Other Study IDs: 2024-07-OSSSZ-6435-LUPELLI
Record Dates: First submitted 2024-10-07; First posted 2024-10-15 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer Surgery; ESPB
Keywords: ESPB

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: ESP block — The ESPB will be performed at the T4 level, monolaterally (according to the surgical side), with 30ml volume of 0.5% Ropivacaine injected with a 20-gauge, 50-mm-long needle. The technique used is the standard ultrasound-guided, sterile procedure.
  Soon after performing the block, a timer will be started to mark the time for subsequent evaluations. At 1,3,5 and after every 5 minutes following the block until 40 minutes or until general anaesthesia is induced, the cold sensitivity of the chest will be explored.

SUMMARY:
The goal of this observational study is to to evaluate the changes in cold sensitivity and the onset of sensory block after performing a thoracic ESP block. It reflects the time it takes for the local anaesthetic to spread into the paravertebral space leading to changes in cold sensitivity in the chest.

The study population are patients undergoing simple quadrantectomy or partial resection with or without sentinel lymphnode removal, in the operating rooms of Santa Maria Goretti Hospital in Latina.

This study is observational because it simply describes and records the effects of a procedure (the ESP block) on treated patients during a period of observation.

Before surgery, unilateral thoracic ESP block (T4 level) with a sterile, ultrasound-guided technique will be performed. A timer will be started to mark the time for subsequent evaluations. At 1,3,5 and after every 5 minutes following the block up to 40 minutes or until induction of general anaesthesia, the cold sensitivity of the chest will be explored.

DETAILED DESCRIPTION:
Breast cancer is the most frequent cancer pathology in women, accounting for 30% of all cancer pathology in women in Italy. Treatment depends on the stage at diagnosis and the histotype, but the surgical approach remains the cornerstone of treatment with radical intent.

Ensuring adequate analgesia during breast surgery can be difficult due to the extensive nature of the surgery and the complex innervation of the breast.

The breast is a subcutaneous organ that receives innervation from the anterior and lateral cutaneous branches of the intercostal nerves T2 to T5 (with varying contributions from T1, T6 and T7) and the supraclavicular nerves from the cervical plexus (C3-C5). The anterior cutaneous branches of the intercostal nerves T2 to T5 cross the pectoralis major muscle near the sternum to innervate the medial quadrants of the breast. The supraclavicular nerves cross the clavicle and innervate the skin below the clavicle and part of the upper pole of the breast. The lateral skin branches of the intercostal nerves from T2 to T5 further divide into anterior and posterior divisions, which perforate the serratus muscle. The anterior divisions provide innervation to the lateral quadrants of the breast. The posterior divisions penetrate the subcutaneous tissue to innervate the lateral thoracic wall. The lateral cutaneous branch of T2 gives rise to the intercostobrachial nerve, which innervates the axilla and the medial upper arm. The first intercostal nerve rarely gives off a lateral cutaneous branch. The lateral and anterior branches of the different intercostal nerves frequently communicate with each other along their course, producing a highly variable pattern of innervation that does not adhere to the rigid dermatomeric segmentation.

Adequate pain control during and after breast surgery improves functional recovery and helps prevent the development of chronic post-operative pain.

Several neuroaxial and regional anaesthesia techniques have been proposed and studied for perioperative pain control.

The paravertebral block (PVB) is considered the gold standard; however it is a complex technique due to its anatomical proximity to the pleura and the central neuroaxial system and is therefore burdened by complications such as pneumothorax and intrathecal local anaesthetic spread.

The erector spinae plane block (ESPB) is a valid alternative to the PVB with characteristics of greater safety and ease of execution but with similar efficacy.

It consists of an ultrasound-guided injection of local anaesthetic (LA) into the virtual fascial plane between the tips of the vertebral transverse processes and the erector spinae muscles.

Depending on the vertebral level chosen, it is indicated for the (uni- or bilateral) analgesia of the thoraco-abdominal wall in various clinical contexts: thoracic surgery, breast surgery, rib fractures, chronic neuropathic pain, abdominal surgery, urological and gynaecological surgery, but also pelvic and knee surgery.

The patient is asked to assume the sitting position; vital parameters are monitored and a thorough skin disinfection is performed. The high-frequency linear probe (5-15 Hz), covered with a sterile sheath, is placed in sagittal paramedian orientation, approximately 2 cm lateral to the spinous process of the fourth thoracic vertebra. It is slid horizontally until the tip of the transverse process is identified and superficially to it the three muscle layers (from surface to depth): trapezius muscle, great rhomboid muscle and the erector muscles of the spine. A 20-gauge, 50-mm-long needle is inserted in plane until it reaches the transverse process, always keeping the structures under ultrasound vision.

After confirming the proper position of the needle tip with the administration of 0.5-1 ml of sterile saline solution, 20-30 ml of local anaesthetic is injected to perform the block. The LA spreads within this virtual plane, up to 3-6 vertebral levels in both cranial and caudal directions; the mediolateral extension is usually confined to the limits of the spinal erector muscle, given by its attachment to the costal angle and the thoracolumbar fascia.

The success of the ESPB mainly depends on a 'paravertebral by proxy' mechanism, i.e. the diffusion of the local anaesthetic in the paravertebral space, through the superior costo-transverse ligaments or through the costo-transverse foramen. In the paravertebral space the LA reaches and wets the spinale nerve roots, determining the effect of the ESPB.

However, it is not known how long it takes for this to occur, i.e. the onset of the blockade and how long the anaesthetic continues to spread in the paravertebral space allowing an increase in the affected dermatomeres is currently unknown in the literature. Knowing this timeframe could be useful and helpful in assessing the minimum time required to ensure adequate onset of analgesia after the technique has been performed.

The aim of the study is to assess the extent of sensory changes, described through altered cold sensitivity, after ESPB at the level of the thoracic skin as time passes. The onset of the sensory changes and the extent of anaesthesia on the thoracic dermatomeres indirectly represent the time required for the LA to reach anteriorly the paravertebral space and wet the spinal nerve roots.

The study population are patients undergoing simple quadrantectomy and partial resection with or without lymphnode resection, in the operating rooms of Santa Maria Goretti Hospital in Latina. Each patient will be enrolled after verification of inclusion/exclusion requirements and collection of written informed consent.

Inclusion criteria are

* Age ≥ 18 years.
* ASA score I-II-III.
* Schedule of breast surgery
* Schedule of ESPB
* Consent to the study Exclusion criteria
* Allergy to local anaesthetics
* Cardiopathies, nephropathies, hepatopathies, central or peripheral neuropathies uncompensated
* Infection at the injection site
* Uncooperative patient
* BMI < 20, > 40
* Difficulty in visualising target structures or the LA spread (failure of technique)
* Pregnancy status

The study has been designed as prospective, single-centre, observational. Perioperative data collection will begin upon patient arrival in the operating room and end at the conclusion of surgery.

The study will end after one year or when the planned sample size is reached. Since this is a prospective observational study of an exploratory nature, there are no previous case histories, and involves no additional risk for patients, there is no need for an a priori sample size calculation. An a priori sample size of 30 patients was therefore established.

Patients who are candidates for breast surgery will undergo a standard anaesthesiological evaluation during which their eligibility for the study will be assessed.

As per the standardised procedure, all patients will be informed about the planned anaesthesia technique and will be asked for informed consent to anaesthesia, pointing out the related anaesthesia risks. Patients will then be asked if they wish to participate in the study. If so, they will be given the consent form for the study, accompanied by a full explanation. If yes, the anaesthetist will ask them to sign the informed consent form for the study. Data collected before surgery are: age, sex, weight, height, BMI, ASA score, comorbidities, surgery history.

On the day of surgery, upon arrival in the operating theatre, the patient will be monitored with electrocardiogram, saturimetry, non-invasive pressure. Management will follow the standard currently applied in the operating room, no changes will be made for the following study.

We briefly describe the usual care of the patient: After premedication with Midazolam 1-2 mg, ESPB will be performed with sterile us-guided technique. The block will be performed at the T4 level, monolaterally, with 30ml volume of 0.5% Ropivacaine. A timer will be started to mark the time for subsequent evaluations. At 1,3,5 and after every 5 minutes after the block until 40 minutes or until general anaesthesia is induced, the cold sensitivity of the chest will be explored. Skin areas where the patient will not perceive the sensation of cold, i.e. anaesthetised skin dermatomeres, will be reported on a schematic template attached to each patient's data collection sheet.

Participation in the study will not lead to changes in clinical practice and all interventions will follow usual care. Procedures will be performed under balanced general anaesthesia or intravenous anaesthesia at the attending anaesthetist'discretion.

This study does not alter commonly used anaesthetic procedures. Therefore, participation in this study will not entail any additional risk for patients and there are no direct benefit associated with it.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* ASA score I-II-III.
* Schedule of breast surgery
* Schedule of ESPB
* Consent to the study

Exclusion Criteria:

* Allergy to local anaesthetics
* Cardiopathies, nephropathies, hepatopathies, central or peripheral neuropathies uncompensated
* Infection at the injection site
* Uncooperative patient
* BMI < 20, > 40
* Difficulty in visualising target structures or the LA spread (failure of technique)
* Pregnancy status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing ESP block for simple quadrantectomy and partial resection with or without lymphnode resection
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
The onset of sensory block after thoracic ESP block after one minute | One minute after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after three minutes | 3 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after five minutes | 5 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after 10 minutes | 10 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after 15 minutes | 15 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after 20 minutes | 20 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after 25 minutes | 25 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after 30 minutes | 30 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after 35 minutes | 35 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.
The onset of sensory block after thoracic ESP block after 40 minutes | 40 minutes after ESPB is performed
  Assessment of the onset, the extent and the evolution, as the time passes by, of sensory changes, described through absent or altered cold sensitivity on the thoracic dermatomeres, after performing thoracic (T4 level) ESPB.

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Santa Maria Goretti, Via Lucia Scaravelli, Latina, Italy, Italy

IPD SHARING:
Plan to Share IPD: Undecided